CLINICAL TRIAL: NCT03069300
Title: The Mechanism of Action of N-acetylcysteine for Reducing the Risk of Infection in Alcoholic Hepatitis
Brief Title: N-ACetylcysteine to Reduce Infection and Mortality for Alcoholic Hepatitis
Acronym: NACAH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14SM2383
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Alcoholic Hepatitis; Infection
MeSH Terms: conditions — Hepatitis, Alcoholic; Infections | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prednisolone+NAC (Experimental): 40mg prednisolone once a day for 28 days and 30 minutes of intravenous NAC at 150mg/kg in 250ml 5% dextrose solution followed by 4 hours of intravenous NAC at 50mg/kg in 500ml 5% dextrose solution, followed by 16 hours of intravenous NAC at 100 mg/kg in 1000ml 5% dextrose solution, followed by 4 days of intravenous NAC at 100mg/kg/day in 1000ml 5% dextrose solution
  Interventions: Drug: N-acetyl cysteine (NAC)
- prednisolone (No Intervention): 40mg prednisolone for 28 days

INTERVENTIONS:
Drug: N-acetyl cysteine (NAC)
  Other Names: NAC
  Arms: prednisolone+NAC

SUMMARY:
Recent data have suggested that monocyte oxidative burst defect is associated with the development of infection in patients with severe alcoholic hepatitis. One report found reduced 28 day mortality in patients treated with N-acetylcysteine combined with prednisolone when compared to prednisolone alone. The current study seeks to reveal whether the mechanism by which NAC reduces susceptibility to infection is through improvement of phagocyte oxidative burst.

DETAILED DESCRIPTION:
Randomised controlled trial, open label.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older
* Clinical alcoholic hepatitis:

  * Serum bilirubin >80umol/L
  * History of alcohol excess (>80g/day male, >60g/day female)
  * Less than 4 weeks since admission to hospital
  * Maddrey's discriminant function (DF) >32
  * Informed consent

Exclusion Criteria:

* Alcohol abstinence of >6 weeks prior to randomisation
* Duration of jaundice >3 months
* Other causes of liver disease including:

  * Evidence of viral hepatitis (hepatitis B or C)
  * Biliary obstruction
  * Hepatocellular carcinoma
* Evidence of current malignancy (except non-melanotic skin cancer)
* Previous entry into the study
* Patients with known hypersensitivity or previous reactions to NAC
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Improvement in monocyte oxidative burst | 24 hours
Improvement in ex vivo monocyte oxidative burst | 5 days

SECONDARY OUTCOMES:
Proportion of patients infected | 28 days
  Infection will be defined in two ways: i. by new/change in intravenous antibiotic prescription and ii. published clinical and microbiological criteria for infection in the setting of liver disease
Proportion of patients infected | 90 days
  Infection will be defined in two ways: i. by new/change in intravenous antibiotic prescription and ii. published clinical and microbiological criteria for infection in the setting of liver disease
Death | 28 days
Death | 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Mark Thursz, MD, Principal Investigator — Imperial College London
Locations (1):
- St Mary's Hospital, Imperial College, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
contact investigators

REFERENCES:
- [Background] Nguyen-Khac E, Thevenot T, Piquet MA, Benferhat S, Goria O, Chatelain D, Tramier B, Dewaele F, Ghrib S, Rudler M, Carbonell N, Tossou H, Bental A, Bernard-Chabert B, Dupas JL; AAH-NAC Study Group. Glucocorticoids plus N-acetylcysteine in severe alcoholic hepatitis. N Engl J Med. 2011 Nov 10;365(19):1781-9. doi: 10.1056/NEJMoa1101214. PMID 22070475
- [Result] Vergis N, Khamri W, Beale K, Sadiq F, Aletrari MO, Moore C, Atkinson SR, Bernsmeier C, Possamai LA, Petts G, Ryan JM, Abeles RD, James S, Foxton M, Hogan B, Foster GR, O'Brien AJ, Ma Y, Shawcross DL, Wendon JA, Antoniades CG, Thursz MR. Defective monocyte oxidative burst predicts infection in alcoholic hepatitis and is associated with reduced expression of NADPH oxidase. Gut. 2017 Mar;66(3):519-529. doi: 10.1136/gutjnl-2015-310378. Epub 2016 Feb 9. PMID 26860769